CLINICAL TRIAL: NCT03308526
Title: Prevailing Microorganisms Causing Neonatal Sepsis in Neonatal Intensive Care Unit (Prospective Study)
Brief Title: Prevailing Microorganisms Causing Neonatal Sepsis in Neonatal Intensive Care Unit (Prospective Study)Prevailing Microorganisms Causing Neonatal Sepsis in Neonatal Intensive Care Unit (Prospective Study)
Acronym: PMCNSINICUPS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gehad Abdelnaser (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Gehad Abdelnaser, Principal invistigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: AssiutUPedia51
Record Dates: First submitted 2017-10-08; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-09

CONDITIONS: Neonatal SEPSIS
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prevailing microorganisms causing neonatal sepsis in neonatal intensive care unit of Assiut University children Hospital Methods prospective study conducted in the neonatal intensive care unit in Assiut university children hospital.

DETAILED DESCRIPTION:
Sepsis remains a leading cause of death in the intensive care units and in all age groups worldwide.sepsis was defined as the host's immune response(systemic inflammatory response syndrome) to injury and/or infectious stimuli in the presence of a known(or strongly suspected) infection .early onset neonatal sepsis occurs in utero or might become infected when exposed to potentially pathogenic bacteria,viruses,or fungi during passage through the birth canal.

ELIGIBILITY:
Inclusion Criteria:

* both preterm and full term neonates
* both early onset and late onset neonatal sepsis

Exclusion Criteria:

* Genetic diseases immunocompromized neonates
* Neonates of diabetic mothers
* Neonates of HIV mothers

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates from age zero to 28 days
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Prevention of neonatal sepsis | From september2017 to september 2018
  Recognition of prevailing microorganisms causing neonatal sepsis in neonatal intensive care units to take preventive measures against it to decrease the incidence of neonatal sepsis